CLINICAL TRIAL: NCT02657590
Title: Documentation of Cardiac Arrhythmias After Open Heart Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ziv Beckerman MD (Other)
Responsible Party: Sponsor-Investigator, Ziv Beckerman MD, cardiac surgeon, Rambam Health Care Campus
Organization: Rambam Health Care Campus (Other)
Other Study IDs: v.01_07.09.2015
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Cardiac Arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims at recording cardiac arrhythmias in patients after open heart surgery. The arrhythmias will be monitored during the entire first postoperative period, till six weeks after surgery.

DETAILED DESCRIPTION:
Approximately 30-50% of patients after cardiac surgery develop cardiac arrhythmias, most often atrial, and most frequently atrial fibrillation (AF).

Various risk factors, inter alia, the type of surgery itself are risk factors. The major additional risk factors for postoperative atrial fibrillation are: age, valvular involvement, length of cardiopulmonary bypass and cross-clamp times.

Postoperative atrial fibrillation is associated with increased length of stay, higher morbidity and mortality including stroke.

Documentation of postopertive atrial fibrillation is well gathered during the postopertive length of stay, but scarce information exists regarding the development and occurence of atrial arrhythmias after the patient's discharge.

Additionally, the various management protocols which exists with regard to postoperative atrial fibrillation, rely on continuous treatment of the patients with amiodarone or various other anti-arrhythmic agents for the initial postoperative period, and the initial first month after discharge.

So far there is not an unambiguous recommendation regarding the duration of treatment required with amiodarone after releasing the patient.

The aim of this study is to document and record cardiac arrhythmias in patients after open-heart surgery within the time window since the release from hospital and up to six weeks after surgery.

Results of the study will allow us to fully characterize postoperative arrhythmias and their risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older.
2. Patients after open-heart surgery (any type of surgery).

Exclusion Criteria:

1. Patients with internal pacemaker.
2. patients with known basic arrhythmia (pre-surgery) or patients who are discharged with some arrhythmias.
3. Patients with low response which it is expected that there will not be able to use the monitoring device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 18 and over who underwent open-heart surgery.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Arrhythmia | 6 weeks
  Documention of arrhythmias in patients after open heart surgery during the six (6) weeks after release

CONTACTS AND LOCATIONS:
Overall Officials: ziv Becerman, MD, Principal Investigator — Rambam Hospital

IPD SHARING:
Plan to Share IPD: Undecided